CLINICAL TRIAL: NCT03606668
Title: Virtual Reality (VR) to Improve Quality of Life in Patients Diagnosed With Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00151
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis; Chronic Pain; Neurological Disorder
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain; Nervous System Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- People with Multiple Sclerosis (PwMS) and Chronic Pain (Experimental): Participants with MS will only be able to receive eight treatment sessions in this study group and will complete their treatment over four weeks. Two treatments sessions must be completed each week (of the four weeks) and separated by at least one day.
  Participants will attend a baseline visit with assessment and training procedures and receive their first treatment immediately after all baseline assessments. Participants will then complete the remaining seven treatment sessions over four weeks. At the final treatment session, participants will repeat assessments. One week following the final treatment session, participants will be asked to return to clinic to complete assessments once more to test cumulative benefits one week following treatment end.
  Interventions: Device: HTC Vive Virtual Reality (VR) system

INTERVENTIONS:
Device: HTC Vive Virtual Reality (VR) system — VR treatment will entail use of computer software designed to immerse participants and engage them in exercises. Software includes virtual painting, walking through vivid and calming settings, solving puzzles, among others.

SUMMARY:
Participants with neurological disorders will be recruited to complete sessions of virtual reality (VR) immersion. VR has been shown to have therapeutic benefit in certain patient populations and requires further clinical study to determine the extent to which VR can be used to rehabilitate and reduce symptom burden. This study seeks to pilot newly developed VR methods and collect preliminary data in order to support research grants and inform larger clinical trials. Additionally, this proposed study will explore the tolerability and preliminary efficacy of Virtual Reality (VR), specifically to determine whether VR can acutely reduce the severity of symptom burden caused by neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years of age
* Has been diagnosed by a clinician as having MS
* Able to commit to the designated period of testing
* Able to understand the informed consent process and provide consent to participate in the study
* Capacity to complete study procedures as determined by screening personnel
* A Brief Pain Inventory interference score of at least 3 or more.
* SDMT Z-Score > -3.0
* WRAT4 Standard Score > or = 85

Exclusion Criteria:

* Visual, auditory, and motor deficits that would prevent full ability to understand study
* Visual, auditory, and motor deficits that would prevent full ability to operate VR equipment
* Uncontrolled epilepsy
* Current diagnosis of vertigo
* Uncontrolled mood disorders
* History of Psychosis or Schizophrenia
* Expanded Disability Status Scale (EDSS) Score greater than 6.5
* Unable to tolerate or manipulate VR treatment procedures (as evidenced by VR capability assessment)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Multiple Sclerosis (PwMS) and Chronic Pain: Participants with MS will only be able to receive eight treatment sessions in this study group and will complete their treatment over four weeks. Two treatments sessions must be completed each week (of the four weeks) and separated by at least one day.
  Participants will attend a baseline visit with assessment and training procedures and receive their first treatment immediately after all baseline assessments. Participants will then complete the remaining seven treatment sessions over four weeks. At the final treatment session, participants will repeat assessments. One week following the final treatment session, participants will be asked to return to clinic to complete assessments once more to test cumulative benefits one week following treatment end.
  HTC Vive Virtual Reality (VR) system: VR treatment will entail use of computer software designed to immerse participants and engage them in exercises. Software includes virtual painting, walking through vivid and calming settings, solving puzzles, among others.
Period: Overall Study
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Started | 20
Completed | 18
Not Completed | 2
Not completed — Screen Failure | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.3757)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity - Short Form 3a Score
Description: PROMIS - Pain Intensity - Short Form 3a consists of 3 questions -- participants report on the intensity of pain experienced in the past 7 days. Each question is scored between 1 (had no pain) to 5 (very severe). The total score range is 3-15; the higher the score, the more intense the pain.
Time Frame: Baseline (Week 1), Treatment End (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 12
score on a scale | 0.42 (1.11)

2. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity - Short Form 3a Score
Description: as for outcome 1
Time Frame: Baseline (Week 1), Study End (Week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 12
score on a scale | 2 (3.56)

3. Secondary Outcome: Change in Neuro-Quality of Life (Neuro-QOL) - Fatigue - Short Form Score
Description: Neuro-QOL - Fatigue - Short Form consists of 8 statements -- participants report on fatigue symptoms experienced in the past 7 days. Each statement is scored 1 (never) to 5 (always). The total score range is 8-40; the higher the score, the more severe the fatigue.
Time Frame: Baseline (Week 1), Treatment End (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 12
score on a scale | 5.5 (10.4)

4. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Related Impairment Score
Description: PROMIS - Sleep Related Impairment consists of 16 items. Participants report on sleep related impairment experienced in the past 7 days. Each statement is scored between 1 (not at all) and 5 (very much). The total score range is 16-80; the higher the score, the higher the level of sleep related impairment.
Time Frame: Baseline (Week 1), Study End (Week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 16
score on a scale | 4 (9.67)

5. Secondary Outcome: Change in PROMIS - Fatigue Score
Description: PROMIS-fatigue short form consists of 8 questions -- participants report on the intensity of fatigue experienced in the past 7 days. Each question is scored between 1 (had no fatigue) to 5 (always). The total score range is 8-40; the higher the score, the more intense the fatigue.
Time Frame: Baseline (Week 1), Treatment End (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 12
score on a scale | 2.25 (6.17)

6. Secondary Outcome: Change in PROMIS - Fatigue Score
Description: as for outcome 5
Time Frame: Baseline (Week 1), Study End (Week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
Number analyzed (Participants) | 16
score on a scale | 3.88 (10.54)

ADVERSE EVENTS:
Time Frame: up to 5 weeks
Arm/Group | People With Multiple Sclerosis (PwMS) and Chronic Pain
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | People With Multiple Sclerosis (PwMS) and Chronic Pain (N=20)
Brief motion sickness (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03606668/Prot_SAP_000.pdf